CLINICAL TRIAL: NCT03336294
Title: Functional Characteristic Properties of Skeletal Muscle Tissue Assessed by P31 Spectroscopy in Young and Older Adults
Acronym: CAMUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/10/159; 2012-A01506-37 (Other: ID-RCB)
Record Dates: First submitted 2014-01-07; First posted 2017-11-08 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Muscle strength; SRM P31; Phosphocreatine
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Old group (Other): Subjects involved in the CAMUS study will perform during the SRM P31 a quadricipital physical task at 70% 1-RM.
  Interventions: Radiation: SRM P31
- Young group (Other): Subjects involved in the CAMUS study will perform during the SRM P31 a quadricipital physical task at 70% 1-RM.
  Interventions: Radiation: SRM P31

INTERVENTIONS:
Radiation: SRM P31 — All the volunteers involved in the CAMUS study will perform during the SRM P31 a quadricipital physical task at 70% 1-RM.

SUMMARY:
P31 nuclear magnetic resonance (RMN) Spectroscopy (SRM P31) has currently being poorly used in the field of sarcopenia.

The aim of the CAMUS study is to investigate the feasibility a protocol of SRM P31 at rest, during and after a standardized physical task. The secondary objective is to compare the metabolism of tyhe skeletal muscle tissue assessed by SRM P31 in young and older individuals. A pilot study, cross-sectional study will be conducted. Ten healthy sedentary 70+ years males and 10 sedentary 25 to 30 years old male will be included.

Level of physical activity, physical performances, will be assessed at baseline. RMN (T1; tractography and SRM P31) will be performed. SRM P31 will be performed at rest, during and after an exhausting muscle task at 70% 1-RM. Feasibility will be judged on the rate of valuable variables recorded (>90%) inorganic phosphate (iP), phosphocreatine (PCr) and isoform of adenosine triphosphate (ATP : alfa, beta, gamma).

ELIGIBILITY:
Inclusion Criteria:

* Old group : 70+ years males
* Young group : 25 to 30 years males
* Sedentary males in the 2 groups
* Informed consent

Exclusion Criteria:

* Contraindication to perform a RMN

Ages: 25 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
SRM P31 assessment | Change of SRM P31 between Before and during a standardized physical task
  Feasibility of a protocol of SRM P31 at rest, during and after a standardized physical task defined by a composite criteria : the rate of valuable variables recorded (>90%) inorganic phosphate (iP), phosphocreatine (PCr) and isoform of ATP (alfa, beta, gamma) on the spectre.
SRM P31 assessment | Change of SRM P31 between during and after a standardized physical task
  Feasibility of a protocol of SRM P31 at rest, during and after a standardized physical task defined by a composite criteria : the rate of valuable variables recorded (>90%) inorganic phosphate (iP), phosphocreatine (PCr) and isoform of ATP (alfa, beta, gamma) on the spectre.

SECONDARY OUTCOMES:
T1; tractography and SRM P31 comparison between young and older sedentary adults | Change between Before and during a standardized physical task
  To compare the RMN (T1; tractography and SRM P31) at rest, during and after an exhausting muscle task at 70% 1-RM between young and older sedentary adults.
T1; tractography and SRM P31 comparison between young and older sedentary adults | Change between during and after a standardized physical task
  To compare the RMN (T1; tractography and SRM P31) at rest, during and after an exhausting muscle task at 70% 1-RM between young and older sedentary adults.

CONTACTS AND LOCATIONS:
Overall Officials: Yves ROLLAND, MD; PHD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rolland Y, Lauwers-Cances V, Cournot M, Nourhashemi F, Reynish W, Riviere D, Vellas B, Grandjean H. Sarcopenia, calf circumference, and physical function of elderly women: a cross-sectional study. J Am Geriatr Soc. 2003 Aug;51(8):1120-4. doi: 10.1046/j.1532-5415.2003.51362.x. PMID 12890076
- [Background] Bourdel-Marchasson I, Joseph PA, Dehail P, Biran M, Faux P, Rainfray M, Emeriau JP, Canioni P, Thiaudiere E. Functional and metabolic early changes in calf muscle occurring during nutritional repletion in malnourished elderly patients. Am J Clin Nutr. 2001 Apr;73(4):832-8. doi: 10.1093/ajcn/73.4.832. PMID 11273861